CLINICAL TRIAL: NCT03168048
Title: Oncologic Therapy Support Via Means of a Dedicated Mobile App - a Prospective Feasibility Evaluation
Brief Title: Oncologic Therapy Support Via Means of a Dedicated Mobile App
Acronym: OPTIMISE-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Nils Nicolay, PD Dr. Dr., PD Dr. Dr. Nils Nicolay, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OPTIMISE-1
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Thoracic Neoplasm; Pelvic Neoplasm; Radiotherapy; Complications; Oncologic Disorders; Breast Cancer; Satisfaction; Quality of Life
Keywords: mobile application; radiotherapy; patient-care; mhealth; follow-up; patient satisfaction; quality of life
MeSH Terms: conditions — Thoracic Neoplasms; Pelvic Neoplasms; Breast Neoplasms; Personal Satisfaction; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Single-center prospective exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile application (Experimental): Patients undergoing radiotherapy will receive additional therapy support by an application installed on a mobile device
  Interventions: Other: mobile application

INTERVENTIONS:
Other: mobile application — Oncologic therapy support by means of a mobile application

SUMMARY:
The present single-center prospective exploratory study, conducted at Heidelberg University Hospital, assesses the feasibility of introducing a concept for additional patient care based on a mobile application for patients undergoing radiotherapy. Patients presenting themselves for the irradiation of thoracic or pelvic tumors will be surveyed regarding general performance, treatment-related Quality of Life (QoL) and symptoms and their need to personally consult a physician on a treatment-daily basis by means of a mobile application. The primary endpoint of feasibility will be reached when 80% of the patients have successfully answered 80% of their respective questions scheduled for each treatment day. Furthermore, treatment-related patient satisfaction and diagnosis-related QoL is assessed by PSQ-18 and EORTC questionnaires at the end of radiotherapy and at the first follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Indication for radiotherapy with potentially curative intent of a primarily thoracic or pelvic target
* Karnofsky performance score (KPS) ≥ 70%,
* Ability to initiate the therapy as an outpatient
* ≥ 18 years of age

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility judged by number of questions answered by each patient on each treatment day | 12-14 weeks
  Feasibility will be reached when 80% of the patients have successfully answered 80% of their respective questions scheduled for each treatment day

SECONDARY OUTCOMES:
Treatment-related patient satisfaction | 12-14 weeks
  Treatment-related patient satisfaction will be assessed after therapy completion by means of the adapted PSQ-18 questionnaire.
Diagnosis-related Quality of Life | 12-14 weeks
  Quality of Life will be assessed at before the start and after the completion of radiotherapy, as well as at first follow-up by means of the EORTC QLQ-C30 questionnaire and the respective diagnosis-related questionnaire modules.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Nicolay, PD Dr. Dr., Principal Investigator — Heidelberg Institute of Radiation Oncology (HIRO)
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, Germany, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Shafie RA, Bougatf N, Sprave T, Weber D, Oetzel D, Machmer T, Huber PE, Debus J, Nicolay NH. Oncologic Therapy Support Via Means of a Dedicated Mobile App (OPTIMISE-1): Protocol for a Prospective Pilot Trial. JMIR Res Protoc. 2018 Mar 6;7(3):e70. doi: 10.2196/resprot.8915. PMID 29510971